CLINICAL TRIAL: NCT02110511
Title: Effects of Bean Form and Digestive Enzyme Availability on Postprandial Responses
Brief Title: Body Responses to Bean Physical Form and "Beano"
Acronym: BFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Megan McCrory, Principal investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 1107011010
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Appetite and Glucose Responses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- alpha-gal & blended lentils (Experimental): 3 capsules of alpha-gal taken with blended lentils
  Interventions: Other: blended lentils
- alpha-gal & whole lentils (Experimental): 3 calpsules of alpha-gal taken with whole lentils
  Interventions: Other: whole lentils
- alpha-gal & no lentils (Experimental): 3 capsules of alpha-gal taken with no lentils control
  Interventions: Other: no lentils
- Placebo & blended lentils (Placebo Comparator): 3 capsules of placebo taken with blended lentils
  Interventions: Other: blended lentils
- Placebo & whole lentils (Placebo Comparator): 3 capsules of placebo taken with whole lentils
  Interventions: Other: whole lentils
- Placebo & no lentils (Placebo Comparator): 3 capsules of placebo taken with no lentils control
  Interventions: Other: no lentils

INTERVENTIONS:
Other: blended lentils — blended lentils burritto breakfast
  Arms: Placebo & blended lentils; alpha-gal & blended lentils
Other: whole lentils — whole lentils breakfast burritto
  Arms: Placebo & whole lentils; alpha-gal & whole lentils
Other: no lentils — No lentils control breakfast burritto
  Arms: Placebo & no lentils; alpha-gal & no lentils

SUMMARY:
The aim of this study is to determine the effects of bean physical form (whole versus blended) and Beano on postprandial responses. The postprandial responses the investigators will examine include blood glucose, appetite, metabolic rate, physical symptoms, and mood. To accomplish this aim the investigators will conduct a randomized, placebo-controlled trial in overweight and obese but otherwise healthy (non-diabetic) men and women

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years old
* Body mass index (BMI) 18.5-40 kg/m2
* Generally healthy
* A non-smoker
* Any ethnicity
* Free of chronic diseases and not taking medications or dietary supplements known to affect energy regulation or appetite

Exclusion Criteria:

* Beano drug label warnings including galactosemia, severe liver or kidney disease, allergies or sensitivities to any of the ingredients in Beano
* Peri and postmenopausal women
* Pregnant or lactating women (currently and within the past 1 year)
* Currently dieting or consuming unusual or a medically prescribed diet
* Net weight loss or gain (>5 lbs) within the last six months
* Consuming 1/2c per day or more of legumes, not including peanuts
* Having taken Beano any time in the past 3 months
* Extreme problems digesting beans
* Fasting glucose >126 mg/dl
* Blood pressure >140/90 mmHg
* Moderate intensity or higher intensity exercise > 6 h/wk
* Predicted energy requirement < 2000 kcal/d or >4000 kcal/d

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Appetite | 3 hours
  Subjects were given an appetite questionnaire to complete at time 0, 20, 40, 60, 120 and 180

SECONDARY OUTCOMES:
Blood glucose | 3 hours
  Finger prick blood were taken at time 0, 20, 40, 60, 120 and 180 for glucose measurement using a glucometer
fasting and postprandial energy expentidure | 4 hours
  Fasting energy expenditure was measured for thirty minutes before meal and beano intervensions were given and at postprandial time points 20, 40, 60, 120 and 180, postprandial energy expenditure was measured for 15 minutes at each time point
gastrointestinal symptoms | 3 hours
  At timepoints 0, 20, 40, 60, 120 and 180, gastroinstinal symptoms were assessed using a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Anguah KO, Wonnell BS, Campbell WW, McCabe GP, McCrory MA. A blended- rather than whole-lentil meal with or without alpha-galactosidase mildly increases healthy adults' appetite but not their glycemic response. J Nutr. 2014 Dec;144(12):1963-9. doi: 10.3945/jn.114.195545. Epub 2014 Oct 8. PMID 25411033